CLINICAL TRIAL: NCT05773846
Title: A Phase 3, Randomized, Double-Blind, Saline Placebo- and Active-Controlled, Multicenter Study to Evaluate the Analgesic Efficacy and Safety of Intra-operative Administration of PRF-110 Following Unilateral Bunionectomy
Brief Title: A Study to Evaluate Analgesic Efficacy and Safety of PRF-110 for Post-surgical Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PainReform LTD (Industry)
Collaborators: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRF-110-103
Record Dates: First submitted 2022-11-01; First posted 2023-03-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Bunion
MeSH Terms: conditions — Bunion | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blind, placebo and active-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Before the start of the study, a computer-generated randomization schedule will be prepared for each site. The randomization codes will be stored in a secured area. Uniquely numbered study medication kits will be assigned to subjects according to the randomization codes.
  Randomization will take place on the day of surgery (Day 1) after performance of baseline assessments. Subjects who continue to meet eligibility criteria will be randomized in a 2:2:1 ratio to 1 of the 3 treatment groups:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PRF-110 (Experimental): PRF-110 3.6% ropivacaine, to be applied into the surgical wound
  Interventions: Drug: Ropivacaine
- Saline .9% (Placebo Comparator): Saline .9%, to b be applied into the surgical wound
  Interventions: Drug: Ropivacaine
- Ropivacaine (Active Comparator): Ropivacaine Hydrochloride 0.5%, up to 10 mL, to be applied into the surgical site
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — A long acting formulation of ropivacaine

SUMMARY:
PRF-110 is a viscous, yellowish clear oily solution of ropivacaine intended for administration into surgical sites to provide post-operative analgesia. The pharmacokinetic profile for PRF-110 suggests that its effect could last up to 72 hours. This is A Phase 3, Randomized, Double-Blind, Saline Placebo- and Active-Controlled, Multicenter Study to Evaluate the Analgesic Efficacy and Safety of Intra-operative Administration of PRF-110 Following Unilateral Bunionectomy

DETAILED DESCRIPTION:
PRF-110 is a unique, sustained-release, oil-based solution formulation of ropivacaine intended for administration into surgical sites for the prevention of postoperative pain. The formulation is designed to have an effect for up to 72 hours. It is postulated that PRF-110 will improve postoperative pain management by providing prolonged pain relief at the surgical site; thereby, reducing the amount of systemic analgesia needed after surgery. The slow, local release of ropivacaine following administration of PRF-110 has been demonstrated in dissolution studies, in postoperative pain studies in animals, in an experimental pain study in human volunteers, and in an open-label Phase 2 hernia repair trial to result in very low plasma concentrations of drug, therefore reducing the probability of systemic adverse events. This is a randomized, double-blind study to evaluate the efficacy and safety of PRF-110 compared with saline placebo and with ropivacaine hydrochloride injection administered intraoperatively in subjects undergoing unilateral bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

Subjects must meet all of the following criteria to be eligible for inclusion into the study:

1. Able to provide written informed consent prior to any study procedures.
2. Able to communicate clearly with the Investigators and study staff.
3. Males and females aged 18 years or older.
4. Scheduled for elective primary unilateral first metatarsal bunionectomy surgery (osteotomy and internal fixation) with no ancillary procedures.
5. Female subjects must be surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or practicing doublebarrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than two months prior to screening and commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study.
6. Negative alcohol breath/saliva test and urine drug screen for drugs of abuse at Screening and at Baseline. Subjects with positive results on the alcohol breath/saliva test or urine drug screen at Screening, and/or prior to surgery, will not be allowed to proceed in the study unless the results can be explained by a current prescription or acceptable over-the-counter medication as determined by the Investigator. Note that for those subjects who test positive for tetrahydrocannabinol (THC), if they are willing to abstain from use or consumption of THC-containing products from Screening thru last Follow-up Visit, they may be allowed to participate in the study.
7. American Society of Anesthesiologists (ASA) Physical Status of I or II (see Appendix, Section 14.1).
8. Body Mass Index (BMI) ≤35.

Exclusion Criteria:

subject will be excluded from the study if any of the following criteria are met:

1. Has clinically significant allergies to an opioid, unless has subsequently tolerated other opioids and, in the opinion of the Investigator, could tolerate a rescue drug containing oxycodone.
2. Has a known or suspected allergy to any local anesthetic or to acetaminophen.
3. Has a known or suspected history of alcohol, opiate or other drug abuse or dependence within 12 months prior to screening.
4. Is unable to refrain from alcohol consumption for a period beginning 24 hours prior to surgery through the end of the 72 -hour evaluation period.
5. Has taken any analgesic or non-opioid pain medication other than acetaminophen (e.g., NSAIDs, cyclooxygenase-2 [COX 2] inhibitors) within 12 hours prior to surgery or any aspirin-containing product within 7 days of the Baseline assessments. Aspirin up to 325 mg once daily for cardiovascular prophylaxis is allowed.
6. Has taken any opioid analgesics or used systemic steroids within 4 days of surgery.
7. Has been using opiates or any non-steroidal anti-inflammatory drug chronically (more than 10 consecutive days) anytime over the past 3 months.
8. Has used antipsychotics or antiepileptics within 30 days prior to surgery. Use of sedatives, hypnotics, antianxiety agents, and antidepressants (other than monoamine oxidase inhibitors [MAOIs]) are allowed if being used for a nonpain indication and at a stable dose within the previous 30 days.
9. Has history of or positive test results for HIV or hepatitis B or C at Screening.
10. Has any history of epilepsy, other than childhood febrile seizures, before the age of 6.
11. Has any history of psychosis, current clinically significant symptomatic psychiatric disorder, or a history of suicide attempt in the past 10 years.
12. Has taken herbal agents or nutraceuticals (e.g., chapparal, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian) during any of the 7 days prior to surgery that could potentially confound the analgesic response in the Investigator's opinion.
13. Has transaminase levels > 2 x ULN, or bilirubin level > 1.5 x ULN (unless Gilbert's syndrome), or estimated glomerular filtration rate (eGFR) < 60 mL/min. Has poorly controlled diabetes with hemoglobin A1c >7.5%.

15. Has any clinically significant condition including an acute or chronic painful physical restrictive condition or any other significant laboratory abnormality that would, in the opinion of the Investigator, confound study assessments or adversely affect subject safety. 16. Has received another investigational drug within 30 days of scheduled surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Measurement of patients pain levels as an indication for the analgesic efficacy of PRF-110 | 72 hours
  The primary objective of this study is to compare the analgesic efficacy of PRF-110 with placebo during the first 72 hours after completion of bunionectomy surgery by measuring pain levels using an 11-point Numerical Rating Scale (NRS)

SECONDARY OUTCOMES:
Measurement of patients pain levels of PRF-110 as compared to ropivacaine hydrochloride | 72 hours
  Measurement of patients pain levels using an 11-point NRS in order to compare the analgesic efficacy of PRF-110 with ropivacaine hydrochloride (0=no pain and 10=worst pain imaginable) (0.5%) injection administered as an infiltration analgesic during the first 72 hours after completion of bunionectomy surgery.
Comparison of opiate use to saline placebo | 72 hours
  To compare post-surgery opioid consumption (in morphine milligram equivalents) over 72 hours for PRF-110 with that of saline placebo.
Comparison of opiate use to ropivacaine HCL injection | 72 hours
  To compare post-surgery opioid consumption through 72 hours for PRF-110 with that of ropivacaine injection.
Percentage of opiate free subjects | 72 hours
  To compare the percentage of subjects who were opioid free through 72 hours post-surgery for PRF-110 compared with that of ropivacaine injection.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Woodland International Research Group, Little Rock, Arkansas
  - Clinical Pharmacology of Miami, Miami, Florida
  - Midwest Clinical Research Center, Dayton, Ohio
  - First Surgical Hospital 4801 Bissonnet Street, Bellaire, Texas
  - Legent Orthopedic Hopital, Carrolton, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No